CLINICAL TRIAL: NCT02236468
Title: Creating Homestead Agriculture for Nutrition and Gender Equity in Burkina Faso
Brief Title: Creating Homestead Agriculture for Nutrition and Gender Equity (CHANGE) in Burkina Faso
Acronym: CHANGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Food Policy Research Institute (Other)
Collaborators: Helen Keller International (Other); Foreign Affairs, Trade and Development, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHANGE BF
Record Dates: First submitted 2014-09-03; First posted 2014-09-10 (Estimated); Last update posted 2016-09-19 (Estimated); Status verified 2016-09

CONDITIONS: Anemia; Growth Retardation
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- new EHFP (Experimental): Group newly participating in an enhanced-homestead food production program including home gardening, poultry rearing and nutrition and health behavior change communication since 2014
  Interventions: Other: Enhanced-Homestead Food Production Program (new)
- old EHFP+WASH (Experimental): Group participating in an enhanced-homestead food production program including home gardening and nutrition and health behavior change communication since 2010 + WASH/malaria behavior change communication since 2014
  Interventions: Other: Enhanced-Homestead Food Production Program (old); Behavioral: WASH/malaria behavior change
- new EHFP+WASH (Other): Group newly participating in an enhanced-homestead food production program including home gardening, poultry rearing and nutrition and health behavior change communication since 2014 + WASH/malaria behavior change communication since 2014
  Interventions: Behavioral: WASH/malaria behavior change; Other: Enhanced-Homestead Food Production Program (new)
- old EHFP+WASH+LNS distribution (Other): Group participating in an enhanced-homestead food production program including home gardening and nutrition and health behavior change communication since 2010 + WASH/malaria behavior change communication and distribution of LNS since 2014
  Interventions: Other: Enhanced-Homestead Food Production Program (old); Behavioral: WASH/malaria behavior change; Dietary Supplement: LNS distribution

INTERVENTIONS:
Other: Enhanced-Homestead Food Production Program (old) — Participation in an enhanced-homestead food production program including home gardening and nutrition and health behavior change communication since 2010
  Arms: old EHFP+WASH; old EHFP+WASH+LNS distribution
Behavioral: WASH/malaria behavior change — WASH/malaria behavior change communication
  Arms: new EHFP+WASH; old EHFP+WASH; old EHFP+WASH+LNS distribution
Dietary Supplement: LNS distribution — Distribution of Nutributter (Fanga Degue) for children
  Arms: old EHFP+WASH+LNS distribution
Other: Enhanced-Homestead Food Production Program (new) — Participation in an enhanced-homestead food production program including home gardening, poultry rearing and nutrition and health behavior change communication since 2014
  Arms: new EHFP; new EHFP+WASH

SUMMARY:
The purpose of this study is to assess the long-term impact of the Enhanced Homestead Food Production Program implemented by HKI on household food security and nutritional status, as well as the impact on including additional interventions (BCC on WASH and malaria prevention, distribution of preventive lipid-based nutrient supplements (LNS)) to children aged 6-24 months old, in addition to the standard E-HFP model.

DETAILED DESCRIPTION:
Over the past twenty years, Helen Keller International (HKI) has implemented its Homestead Food Production (HFP) program to increase household production of micronutrient-rich foods and improve the quality of diets among vulnerable households across Asia and, more recently, Africa. As part of the program, village model farms -which support diversified, year-round production of micronutrient-rich crops, and improved breeds of poultry and small animals-are established to demonstrate gardening and small animal-raising techniques to program participants. Program participants in turn are established to demonstrate gardening and small animal-raising techniques to program participants. Program participants in turn are provided with small inputs such as seeds, seedlings, and small tools to establish home gardens using techniques they learn at the village model farms. In addition, the program uses a behavior change communication (BCC) strategy to increase participant's health and nutrition-related knowledge and practices.

In 2010, HKI introduced an enhanced-HFP (E-HFP) model in the Gourma province of Burkina Faso with support from the USAID. The project used a randomized cluster design to assess the impact of HKI's package of interventions on 1,200 beneficiary and 800 control children aged 3-12 months at baseline. Given the encouraging results of IFPRI's first evaluation of that project, HKI is working to continue to improve and evaluate its E-HFP program in Burkina Faso. Based on the recommendations from the initial evaluation in Burkina Faso, this research aims to assess both the long-term impact of the E-HFP program as well as the impact of including additional interventions, using the E-HFP platform to deliver these interventions. The primary research questions that will be addresses will be:

* What is the relative impact of a long-term E-HFP program compared to a short-term E-HFP program on household food security and child nutritional status?
* What is the impact of including additional messages and the promotion of practices related to water, sanitation, hygiene, and malaria prevention (including bednet utilization) in the BCC strategy, in addition to the standard E-HFP model?
* What is the impact of distributing preventive lipid-based nutrient supplements (LNS) to children between the ages of 6-24 months in addition to participation in the E-HFP program + additional messages and the promotion of practices related to water, sanitation, hygiene, and malaria prevention (including bednet utilization)?

ELIGIBILITY:
Inclusion Criteria:

* Mother of child between the ages of 0 and 12 months and her child

Exclusion Criteria:

* N/A

Max Age: 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2747 (Actual)
Dates: Start 2014-03; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Hemoglobin (g/dl) | Measurements will be made for children between the ages of 0 and 12 months of age at baseline and 2 years later, at endline, when the children are between the ages of 24 and 36 months.
  Changes in hemoglobin (g/dl) and in prevalence of anemia (<11g/dl) will be measured over the course of the two year program period.

SECONDARY OUTCOMES:
Dietary diversity (%) | Baseline (2014) and after 24 months at Endline (2016)
  Measured with a questionnaire using a qualitative 24h recall. Unit: Number of food group consumed and percentage of children having consumed 4 groups (upon 7) the previous day .
Food security (%) | Baseline (2014) and after 24 months at Endline (2016)
  Measured with a questionnaire to calculate the HFIAS score. Unit: percentage of household
Biochemical markers | Baseline (2014) and after 24 months at Endline (2016)
  Change in plasmatic concentration of iron biomarkers (tranferrin receptors and ferritin; TfR in mg/L and F in μg/L), in concentration of vitamine A biomarkers (retinolbindingprotein; RBP in μmol/L) and inflammatory proteins (C-reactiveprotein and alpha-1 acidglycoprotein; CRP in mg/L and AGP in g/L).
Women's empowerment (%) | Baseline (2014) and after 24 months at Endline (2016)
  Measured by questionnaire, using a decision-making module and a domestic violence module. Percentage of women over a calculated score.
Maternal health and nutrition/WASH/malaria-related knowledge (%) | Baseline (2014) and after 24 months at Endline (2016)
  Using questionnaire on knowledge. Percentage of women giving adequate answer.
IYCF/WASH/malaria practices (%) | Baseline (2014) and after 24 months at Endline (2016)
  Using questionnaire on practices. Percentage of women with adequate practices.
Growth (Z-score and %) | Measurements will be made for children between the ages of 0 and 12 months of age at baseline and 2 years later, at endline, when the children are between the ages of 24 and 36 months.
  Change in heigh-for-age Z-scores, weight-for-age Z-scores and weight-for-height Z-scores will be measured as well as the change in the prevalence of stunting (HAZ<-2), underweight (WAS<-2) and wasting (WHZ<-2) over the course of the two year program period.

CONTACTS AND LOCATIONS:
Overall Officials: Deanna Olney, PhD, Principal Investigator — International Food Policy Research Institute
Locations (1):
- Hellen Keller International, Fada, Gourma, Burkina Faso